CLINICAL TRIAL: NCT02498509
Title: A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Concomitant Mometasone Furoate and Levocabastine HCl in Perennial Allergic Rhinitis Patients
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-342
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 153PAR14017
Record Dates: First submitted 2015-07-05; First posted 2015-07-15 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2015-07

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Mometasone Furoate; levocabastine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment (Experimental): CKD-342
  Interventions: Drug: CKD-342
- Control 1 (Active Comparator): Mometasone furoate
  Interventions: Drug: Mometasone furoate
- Control 2 (Active Comparator): Levocabastine HCL
  Interventions: Drug: Levocabastine HCL

INTERVENTIONS:
Drug: CKD-342 — treatment for 4 weeks after randomization
  Other Names: investigational product
  Arms: Treatment
Drug: Mometasone furoate — treatment for 4 weeks after randomization
  Other Names: investigational product
  Arms: Control 1
Drug: Levocabastine HCL — treatment for 4 weeks after randomization
  Other Names: investigational product
  Arms: Control 2

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of CKD-342

DETAILED DESCRIPTION:
A Randomized, Double-blind, Active-controlled, Multicenter phase 3 Clinical trial to evaluate the Efficacy and Safety of Concomitant Mometasone furoate and Levocabastine HCl in Perennial Allergic Rhinitis patients

ELIGIBILITY:
Inclusion Criteria:

1. male, female, Age: over 13 years(no age limiation in upper)
2. subject who has experienced perennial allergic rhinitis for over 1 year
3. subject who has identified allergens throughout the year within 12 months
4. subject who has the symptoms of moderate to severe allergic rhinitis
5. subject who can record the the patient diary during the clinical trial period
6. subject who agreed to keep the same environment during the clinical trial period

Exclusion Criteria:

1. Asthma
2. Previous medical history at screening (Nasal polyps within the previous two months, biopsies, ulcers, trauma, surgery, atrophic rhinitis, patients with a history of drug rhinitis)
3. Patients with untreated localized infection in nasal mucosa
4. Patients following administration of a combination of prohibited drugs in patients administered concomitant medications or trial period is expected to be inevitable
5. Patients with abnormal following laboratory test results at screening

   * AST, ALT>2times the upper limit of normal at screening
   * Serum creatinine >1.5times the upper limit of normal at screening
6. Previous history of acute or severe chronic sinusitis within 30 days at screening
7. The continue use of drugs that may affect the efficacy of the Investigational product
8. Start the immunotherapy or a change of doge within 1 month, at screening
9. If you have glaucoma or cataracts, herpes simplex, or around the eyes
10. Chronic obstructive pulmonary disease (COPD)
11. history of hypersensitivity reactions and for treaties or major components of the IP
12. Pregnant women, breast feeding women or women of childbearing potential must agree to use appropriate contraception methods
13. Alcohol or illegal drug abuse or dependence in patients
14. participation in any investigational or maketed drug within 4weeks preceding the screening visit
15. Patients that can not be participating in a clinical trial by investigator's discretion

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
change in rTNSS from baseline | up to week 4

SECONDARY OUTCOMES:
change in rTNSS from baseline | up to week 2
change in AM rTNSS and PM rTNSS from baseline | 2 weeks and 4 weeks after the baseline assessment
Physician assessed overall nasal symptom from baseline | 2 weeks and 4 weeks after the basline assessment
change from baseline in RQLQ | 2 weeks and 4 weeks after the baseline assessment
Changing in 4 nasal symptom score (sneezing, runny nose, nasal congestion, itchy nose) from baseline | 2 weeks and 4 weeks after the basline assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Irwon-dong, Gangnam-gu, Seoul, South Korea